CLINICAL TRIAL: NCT02852018
Title: Identification of Genetic Markers Modulating Rhythmic Risk Among Patients With Severe Cardiomyopathy
Acronym: GENECHOC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/10/77
Record Dates: First submitted 2016-07-21; First posted 2016-08-02 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Appropriate treatment: Patients who have a rhythmic event (before or after inclusion) appropriately treated either by administering an electric shock or by antiarrhythmic stimulation
  Interventions: Genetic: Identification of genetic polymorphisms
- No event: Patients who have never received treatment or electrical antiarrhythmic stimulation and with a minimum follow-up of three years before inclusion and did not receive appropriate treatment during the follow up period of the study.
  Interventions: Genetic: Identification of genetic polymorphisms

INTERVENTIONS:
Genetic: Identification of genetic polymorphisms

SUMMARY:
The aim of this project is to identify common genetic polymorphisms associated with the occurrence of rhythmic events in patients with severe cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted for primary prevention, an implantable cardioverter defibrillator (ICD) single or double room, for severe cardiomyopathy (EF <35%)
* Patients with ischemic cardiomyopathy or idiopathic dilated cardiomyopathy.- "Appropriate treatment" group: patients who had a rhythmic event (before or after inclusion) appropriately treated either by administering an electric shock or by antiarrhythmic stimulation
* Group "no event" patients who have never received treatment or electrical antiarrhythmic stimulation and with a minimum follow-up of three years before inclusion and did not receive proper treatment during the follow up period of the study

Exclusion Criteria:

* Patients implanted with an ICD for primary prevention in the context of a family hereditary disease (long QT syndrome, Brugada syndrome, hypertrophic cardiomyopathy, ventricular tachycardia catecholergic right ventricular dysplasia ...).
* Patients with left ventricular function greater than 35%.
* Patients implanted with a defibrillator function resynchronization.
* Patients minors, adults under guardianship and protected persons are eligible under this project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Genetic analysis will compare 500 patients implanted with an ICD for primary prevention and having received an appropriate shock and another 500 patients implanted with an ICD for primary prevention and have not received appropriate shock after a minimum follow-up three years before inclusion. To allow the matching of two groups, it requires to recruit 500 patients in the "appropriate treatment" group and 1000 patients in the "no event" group.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of polymorphisms pre-selected candidates (or by direct sequencing by High Resolution Melting). | 4 years
Identification of polymorphisms frequent (> 5% in the general population) by association study ( "Genome Wide Association Study '(GWAS)) using genotyping technology broadband Axiom (Affymetrix). | 4 years

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Clermont-Ferrand., Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CH La Rochelle, La Rochelle
  - CHRU Lille, Lille
  - CHU Lyon, Lyon
  - CHU Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No